CLINICAL TRIAL: NCT00615745
Title: A Phase IV, Open-label, Prospective Observational Study to Evaluate Virological Response in Antiretroviral-Experienced HIV 1 Infected Subjects Switching to Atripla (Efavirenz/Emtricitabine/Tenofovir DF) on an Empty Stomach
Brief Title: ONCE - Only Nocturnal Combination Evaluation of Antiretroviral-Experienced HIV 1 Infected Subjects Switching to Atripla
Acronym: ONCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-EU-177-0111; EudraCT Number 2007-005769-36
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Atripla (ATR) consisting of EFV 600 mg/FTC 200 mg/TDF 300 mg as one tablet orally once daily taken on an empty stomach at bedtime.
  Interventions: Drug: Atripla (ATR) consisting of EFV 600 mg/FTC 200 mg/TDF 300 mg

INTERVENTIONS:
Drug: Atripla (ATR) consisting of EFV 600 mg/FTC 200 mg/TDF 300 mg — Atripla (ATR) consisting of EFV 600 mg/FTC 200 mg/TDF 300 mg as one tablet orally once daily taken on an empty stomach at bedtime.

SUMMARY:
A single tablet regimen (STR) of efavirenz, emtricitabine and tenofovir disoproxil fumarate (tenofovir DF) is the first complete HAART that is offered as one tablet once a day. The individual components of this HAART regimen have demonstrated efficacy and safety in HIV treatment-naive patients and offer simplification that in turn may increase adherence and improve clinical outcomes. This study aims to evaluate the effectiveness (efficacy, safety and tolerability) of a STR simplification strategy in patients on HAART who have achieved viral suppression in a real world clinical setting.

DETAILED DESCRIPTION:
This is a prospective study to evaluate pure virological response rates in antiretroviral-experienced HIV infected subjects initiating therapy with Atripla. Subjects will be switching to Atripla having already been established on the individual components of efavirenz, emtricitabine, and tenofovir DF.

Within the Chelsea and Westminster hospital approximately 540 subjects have been identified who are currently receiving the individual components of Atripla and who would eventually switch to Atripla. The Royal Sussex County Hospital will be included to ensure that recruitment timelines are met.

A minimum of 150 subjects will be switched within the first 6 months allowing initial 24 week data for these subjects to be available approximately 12 months post launch.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have documented HIV 1 infection by Roche Amplicor (Version 1.5 Ultra sensitive) or equivalent assay - either at screening or previously documented in the patient's medical record.
* Stable HAART regimen of efavirenz, emtricitabine and tenofovir DF for equal to or greater than 24 weeks prior to Screening and must be on their first HAART regimen.
* Undetectable plasma HIV 1 RNA (less than 50 copies/mL) at Screening and greater than or equal to 12 weeks prior to Screening.
* Greater than or equal to 18 years old.
* Adequate renal function by: Estimated creatinine clearance greater than or equal to 60 mL/min according to the Cockcroft Gault formula
* Hepatic transaminases (AST and ALT) less than or equal to 5 times upper limit of normal (ULN)
* Total bilirubin less than or equal to 1.5 mg/dL
* Adequate hematologic function (absolute neutrophil count greater than or equal to 1,000/mm3; platelets greater than or equal to 25,000/mm3; hemoglobin greater than or equal to 8.0 g/dL
* Serum amylase less than or equal to 1.5 times ULN (subjects with serum amylase greater than 1.5 times ULN will remain eligible if serum lipase is less than or equal to 1.5 times ULN)
* Negative serum pregnancy test (females of childbearing potential only i.e., not surgically sterile or at least two years post-menopausal)
* Women of childbearing potential (WOCBP) must be willing to use two methods of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drugs in such a manner that the risk of pregnancy is minimized. Subjects may choose two (a barrier and highly effective method) of the birth control methods listed below: Hormonal birth control drugs, Male or female condoms with or without spermicidal gels, Diaphragm cervical cap with or without spermicidal gels, Intrauterine device
* Female subjects who utilize hormone contraceptive as one of their birth control methods must have used the same methods for at least three months prior to study dosing.
* Female subjects who are postmenopausal for less than two years are required to have FSH greater than or equal to 40 mIU/mL. If the FSH is less than 40 mIU/mL, the subject must agree to use highly effective method of birth control (as described above) to participate in the study.
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condom with spermicide) during heterosexual intercourse from screening through completion of the study and continuing for up to 12 weeks after the last dose of study drugs.
* Life expectancy greater than or equal to 1 year.
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* Known hypersensitivity or toxicities to emtricitabine (FTC), tenofovir DF (TDF) or Truvada
* Known hypersensitivity or toxicities to Sustiva
* Have a history of resistance to any of the study agents at the time of screening (documented presence of resistance mutation(s) as defined by the IAS-USA 2007 Guidelines
* A new AIDS-defining condition diagnosed within the 30 days prior to the Baseline visit.
* Pregnant/lactating or breastfeeding females
* Severe hepatic impairment (greater than 5 times upper limit of normal as defined by laboratory transaminases) or deemed clinically significant by investigator.
* Any currently known clinical or laboratory parameter of GSI Grade 4. However asymptomatic grade 4 abnormalities will be permitted at the discretion of the investigator if deemed clinically appropriate (excluding AEs and laboratory parameters mentioned elsewhere in the inclusion/exclusion criteria). Abnormalities deemed insignificant by the investigator must be discussed with the sponsor prior to enrollment.
* Receiving on-going therapy with any of the prohibited medications. Administration of any of the medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period.
* Active, serious infections (other than HIV infection) requiring parenteral antibiotic therapy within 30 days prior to Screening visit.
* Current acute illness or infection (e.g., opportunistic) - including an active AIDS defining condition within the previous six months.
* Hepatitis B coinfection or Hepatitis C coinfection
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Subjects with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS with 30 days of Baseline visit and are not anticipated to require systemic therapy during the study.
* Prior history of renal or bone disease deemed significant by the investigator.
* Subjects currently taking part in any other clinical trial using an investigational product, with the exception of studies where the treatment studied has been stopped for more than 1 month.
* Evidence of alcohol and/or drug or substance abuse that in the judgment of the investigator would likely result in the patient being unreliable in fulfilling the conditions of the protocol.
* History of psychological illness or conditions that in the judgment of the investigator might interfere with the patient's ability to understand the requirements of the study.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements and cause the patient to be unable to complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of subjects who maintain pure virologic response at HIV 1 RNA threshold of 50 copies/mL (PVR50; lack of confirmed HIV 1 RNA level greater or equal to 50 copies/mL) through Week 48. | 48 weeks

SECONDARY OUTCOMES:
Proportion of subjects who have pure virologic response at HIV 1 RNA threshold of 400 copies/mL (PVR400; lack of confirmed HIV 1 RNA level greater or equal to 400 copies/mL) through Week 48. | 48 weeks
Proportion of subjects who have PVR50 at Week 24. | 24 weeks
Proportion of subjects who have PVR400 at Week 24. | 24 weeks
Change from baseline in CD4 cell count through 48 weeks of treatment. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cham Herath, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Cambridge, United Kingdom